CLINICAL TRIAL: NCT06820853
Title: Single-shot Versus Slow Infusion Interscalene Block and Its Impact on Diaphragmatic Function in Patients Undergoing Shoulder Surgery, a Randomized Controlled Trial
Brief Title: Single-shot Versus Slow Infusion Interscalene Block and Its Impact on Diaphragmatic Function in Patients Undergoing Shoulder Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: interscalane block and DE
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-02

CONDITIONS: Brachial Plexus Blockade

STUDY DESIGN:
Intervention Model Description: patients will be randomly allocated into 2 groups : single shot group and slow infusion group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single shot (Active Comparator): They will receive a 10 ml of 0.5 % bupivacaine as a single shot
  Interventions: Device: Diaphragmatic excursion evaluation
- Slow administration group (Active Comparator): They will receive 10 ml of 0.5% bupivacaine over 10 minutes
  Interventions: Device: Diaphragmatic excursion evaluation

INTERVENTIONS:
Device: Diaphragmatic excursion evaluation — They will receive 10 ml of 0.5% bupivacaine over 10 minutes

SUMMARY:
Interscalene brachial plexus block is a commonly chosen anesthetic technique for shoulder and proximal arm surgery yet it carry several risks including phrenic nerve block.

Researchers assumed that slow administration of local anesthetic would reduce incidence of phrenic nerve block

DETAILED DESCRIPTION:
patients will be randomly allocated into one of 2 groups ( single shot group) and slow administration group . single shot will receive a 10 ml bolus of 0.5% bupivacaine the other group will receive 10 ml 0.5 % bupivacaine over 10 minutes (at a rate of 1ml/minute) using syringe pump An experienced operator who will be blinded to method of administration will conducted diaphragmatic excursion of ipsilateral hemidiaphragm using curved probe at baseline and at 10 minutes interval for 30 minutes Complete phrenic will be defined as 75% or more reduction in DE, while partial failure as 25%-50% reduction in DE

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II undergoing shoulder surgery under GA

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Complete phrenic nerve block defined as > 75% reduction in diaphragmatic excursion | baseline and 30 minutes after the block
  defined as > 75% reduction in diaphragmatic excursion

SECONDARY OUTCOMES:
partial phrenic block | baseline and 30 minutes after the block
  25-50% reduction in DE

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from corresponding author upon reasonable request

REFERENCES:
- [Background] Renes SH, Rettig HC, Gielen MJ, Wilder-Smith OH, van Geffen GJ. Ultrasound-guided low-dose interscalene brachial plexus block reduces the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):498-502. doi: 10.1097/AAP.0b013e3181b49256. PMID 19920426
- [Background] Wong AK, Keeney LG, Chen L, Williams R, Liu J, Elkassabany NM. Effect of Local Anesthetic Concentration (0.2% vs 0.1% Ropivacaine) on Pulmonary Function, and Analgesia After Ultrasound-Guided Interscalene Brachial Plexus Block: A Randomized Controlled Study. Pain Med. 2016 Dec;17(12):2397-2403. doi: 10.1093/pm/pnw057. Epub 2016 Apr 13. PMID 28025374
- [Background] Fujimura N, Namba H, Tsunoda K, Kawamata T, Taki K, Igarasi M, Namiki A. Effect of hemidiaphragmatic paresis caused by interscalene brachial plexus block on breathing pattern, chest wall mechanics, and arterial blood gases. Anesth Analg. 1995 Nov;81(5):962-6. doi: 10.1097/00000539-199511000-00012. PMID 7486085
- [Background] Verelst P, van Zundert A. Incidence of phrenic nerve block after interscalene brachial plexus block. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):411-2; author reply 412. doi: 10.1097/AAP.0b013e318219e19d. No abstract available. PMID 21697691
- [Background] Mitchell C, Adebajo A, Hay E, Carr A. Shoulder pain: diagnosis and management in primary care. BMJ. 2005 Nov 12;331(7525):1124-8. doi: 10.1136/bmj.331.7525.1124. No abstract available. PMID 16282408
- [Background] Urwin M, Symmons D, Allison T, Brammah T, Busby H, Roxby M, Simmons A, Williams G. Estimating the burden of musculoskeletal disorders in the community: the comparative prevalence of symptoms at different anatomical sites, and the relation to social deprivation. Ann Rheum Dis. 1998 Nov;57(11):649-55. doi: 10.1136/ard.57.11.649. PMID 9924205
- [Derived] Helmy MA, Gamal B, Milad LM, Adawy AE, Ibrahium F, Kasem S, Mustafa H. Single-shot versus slow infusion interscalene block and its impact on diaphragmatic function in patients undergoing shoulder surgery, a double blind randomized controlled trial. Anaesth Crit Care Pain Med. 2025 Nov 7:101668. doi: 10.1016/j.accpm.2025.101668. Online ahead of print. PMID 41207378